CLINICAL TRIAL: NCT06308523
Title: A Randomized, Double-blind, Placebo-controlled Multiple-ascending Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AP303 Following 2-week Oral Administration in Healthy Chinese Participants.
Brief Title: A Study to Evaluate the Safety, Tolerability, PK and PD of AP303 in Healthy Chinese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alebund Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AP303-PK-02
Record Dates: First submitted 2024-02-20; First posted 2024-03-13 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AP303 (Experimental)
  Interventions: Drug: AP303 150 μg; Drug: AP303 300 μg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo 150 μg; Drug: Placebo 300 μg

INTERVENTIONS:
Drug: AP303 150 μg — AP303 Tablet 150 μg QD
  Arms: AP303
Drug: Placebo 150 μg — Placebo Tablet 150 μg QD
  Arms: Placebo
Drug: AP303 300 μg — AP303 Tablet 300 μg QD
  Arms: AP303
Drug: Placebo 300 μg — Placebo Tablet 300 μg QD
  Arms: Placebo

SUMMARY:
The study will be a single center, double-blind, randomized, placebo-controlled, multiple-ascending-dose study to evaluate the safety, tolerability, PK and PD of AP303 following 2-week oral administration to healthy Chinese participants.

DETAILED DESCRIPTION:
Eligible study participants will be enrolled and randomized into one of the two dose cohorts, each cohort will include 9 participants randomized to AP303 and placebo at 2:1 ratio (6 on AP303 and 3 on placebo).

ELIGIBILITY:
Important Inclusion Criteria:

1. Healthy male and female participants, 18-50 years of age.
2. BMI (body mass index) 18-27 kg/m2.

Important Exclusion criteria:

1. History or symptoms of any clinically significant kidney, liver, broncho-pulmonary, gastrointestinal, neurological, psychiatric, cardiovascular, endocrine/metabolic, hematological disease or cancer.
2. Personal history of congenital long QT syndrome or family history of sudden death.
3. People with a history of specific severe allergies, or severe allergic conditions or known allergies to the study or any of its ingredients or excipients as judged by the investigator, or any acute confirmed significant allergic reactions to any drug, or multiple drug severe allergies (non-active hay fever is acceptable). Allowing for childhood asthma, history of mild eczema that has had no flare ups for ≥5 years or is fully resolved.
4. History of having received or currently receiving any systemic anti-neoplastic or immunomodulatory treatment (including systemic oral or inhaled corticosteroids) ≤6 months prior to the first dose of study drug or the expectation that such treatment will be needed at any time during the study.
5. Participants who have had significant acute infection, e.g., COVID-19, influenza, local infection, acute gastrointestinal symptoms or any other clinically significant illness within two weeks before study drug administration.
6. Confirmed systolic BP greater than 140 or less than 90 mmHg, and diastolic BP greater than 90 or less than 50 mmHg at screening.
7. Abnormalities of ECG parameters and abnormal shape of ECG wave on screening ECG.
8. Implantation of cardiac pacemaker or clinically significant arrhythmias.
9. Estimated glomerular filtration rate (eGFR) <90 mL/min/1.73 m2 (using the CKD-EPI equation).
10. Positive test at screening of any of the following: Hepatitis B (HBsAg), Hepatitis C (HCVAb), human immunodeficiency virus (HIV Ab) or syphilis AB.
11. ALT or AST >1.5 × ULN, or any other clinically significant abnormalities in laboratory test results at screening.
12. Dosed with a small-molecule or biologic investigational drug within 30 days or 90 days, respectively, or 5 half-lives whichever is the longer) prior to first dose of this study.
13. Donation of component (plasma or platelet) or whole blood ≥200 mL within 4 weeks prior to screening.
14. Receipt of a live vaccine within 4 weeks of prior to screening (Influenza and COVID-19 vaccines are allowed).
15. Positive urine test for drugs of abus.
16. History of drug and/or alcohol abuse or addiction.
17. History (within 3 months of screening) of alcohol consumption exceeding 2 standard drinks per day on average (1 standard drink = 10 grams of alcohol). Alcohol consumption within 48 hours before screening.
18. Use of >5 cigarettes or equivalent nicotine-containing product per day.
19. Taking any prescribed or over-the-counter medications (including vitamins or herbal remedies) within 30 days or 5 half-lives (whichever is the longer) of the first dose of study drug. Occasional paracetamol is allowed (see section on Permitted Therapy). Exceptions may be made on a case-by-case basis following discussion and agreement between the investigator and the sponsor.
20. Medical or social conditions that would potentially interfere with the participant's ability to comply with the study visit schedule or the study assessments.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2024-03-18 (Actual); Primary Completion 2024-05-13 (Actual); Study Completion 2024-05-13 (Actual)

PRIMARY OUTCOMES:
Cmax | Day 1, Day 3-14
  Maximum observed plasma concentration
Tmax | Day 1, Day 3-14
  Time to maximum observed plasma concentration
AUC0-24h | Day 1
  Area under the plasma concentration versus time curve up to 24 hours
AUC0-last | Day 1
  Area under the plasma concentration versus time curve up to the last measurable concentration
AUC0-inf | Day 1
  Area under the plasma concentration versus time curve extrapolated to infinity
AUC0-t | Day 3-14
  Area under the plasma concentration-time curve for a dosing interval
t1/2 | Day 1, Day 3-14
  Apparent terminal half-life, computed as ln(2)/λz
CL/F | Day 1
  Apparent oral clearance calculated from Dose/ AUC0-inf
V/F | Day 1, Day 3-14
  Apparent volume of distribution of oral drug
Cav | Day 3-14
  average plasma concentration
Ctrough | Day 3-14
  Trough plasma concentration
Rac | Day 3-14
  Ratio of accumulation
Incidence and severity of adverse events | Day 1-28
  Incidence and severity of adverse events
Incidence of laboratory abnormalities, based on hematology, clinical chemistry, coagulation and urinalysis test results | Day 1-28
  Incidence of laboratory abnormalities, based on hematology, clinical chemistry, coagulation and urinalysis test results
Effect of AP303 on ECG parameters | Day 1-28
  Heart rate in beats/min
Effect of AP303 on ECG parameters | Day 1-28
  QT in ms
Effect of AP303 on ECG parameters | Day 1-28
  PR in ms
Effect of AP303 on ECG parameters | Day 1-28
  QRS in ms
Effect of AP303 on ECG parameters | Day 1-28
  QTcF in ms
Effect of AP303 on ECG parameters | Day 1-28
  QTcB in ms
Vital signs | Day 1-28
  Effect of AP303 on vital signs, e.g. blood pressure
Effect of AP303 on physical examination result | Day 1-28
  nature, frequency, and severity of abnormality of physical examination result
body weight | Day 1-28
  Effect of AP303 on body weight, e.g. change of body weight after administration of AP303

SECONDARY OUTCOMES:
Fasting glucose | Baseline, Days 5, 10, 14 and 28
  Fasting glucose
Fasting lipid profile | Baseline, Days 5, 10, 14 and 28
  Triglyceride, HDL-C, LDL-C, Total cholesterol
Serum creatinine | Baseline, Days 5, 10, 14 and 28
  Serum creatinine
eGFR | Baseline, Days 5, 10, 14 and 28
  Estimated glomerular filtration rate

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No